CLINICAL TRIAL: NCT01306552
Title: BEST Prevention Study. "Berlin Evaluates School Tabacco Prevention" Study Evaluation of a Combined Parent-student Programme for Smoking Prevention in Berlin Schools
Brief Title: Evaluation of a Combined Parent-student Programme for Smoking Prevention in Berlin Schools
Acronym: BEST
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: Senatsverwaltung für Bildung, Wissenschaft und Forschung, Berlin, Germany (Unknown); KARUNA prevents, Berlin, Germany (Unknown)
Responsible Party: Prof. Dr. Stefan N. Willich, Director, Institute for Social Medicine, Epidemiology and Health Economics, Charité University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: EA1/133/10
Record Dates: First submitted 2011-03-01; First posted 2011-03-02 (Estimated); Last update posted 2011-03-02 (Estimated); Status verified 2011-01

CONDITIONS: Tobacco Use Disorder
Keywords: Tobacco use; Adolescents; Primary prevention; Program effectiveness; Parental component
MeSH Terms: conditions — Tobacco Use Disorder; Tobacco Use | interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Student-intervention only group (Active Comparator): Schools randomized to intervention only (arm 1) will agree to visit the smoking prevention parcours offered by KARUNA e.V. ("Rauchst Du noch oder lebst Du schon?").
  One school class of students will visit the parcours once during a school day. The parcours takes approximately 3 hours to complete. The parcours consists of 7 interactive stations where a class of students learns about differences between smokers and non-smokers in terms of health status such as atherosclerosis prevalence, loss of smell or lung capacity and aging. Students also learn about the toxic ingredients in cigarettes. Each station includes a quiz to complete by each group of students. At the end of the parcours, a moderator will announce which group of students accumulated the most points. For more information on the contents of the parcours see http://www.karuna-prevents.de/index.php.
  Interventions: Behavioral: Student-Intervention only group
- Multi-component intervention (Active Comparator): Schools randomized to the student-parent intervention arm also will agree to visit the KARUNA e.V. smoking prevention parcours. In addition, the schools will agree to have one parents' night presented by trained health coaches informing parents about smoking prevention topics in youth during the school year. Trained health coaches will give an evaluated smoking prevention presentation for parents at the parents' nights at the end of the first school year. Also, participating parents will receive information about successful ways to prevent smoking and promote smoking cessation in their children once by mail.
  Interventions: Behavioral: Multi-component Intervention
- Control Group (Active Comparator): Schools randomized to the control school will be offered to participate in the nutrition and exercise prevention program offered by KARUNA e.V. during the 2-year study.
  Interventions: Behavioral: Control Group

INTERVENTIONS:
Behavioral: Student-Intervention only group — One visit to the smoking prevention parcours offered by KARUNA e.V. ("Rauchst Du noch oder lebst Du schon?") during 7th grade.
  The parcours takes approximately 3 hours to complete. The parcours consists of 7 interactive stations where a class of students learns about differences between smokers and non-smokers in terms of health status such as atherosclerosis prevalence, loss of smell or lung capacity and aging. Students also learn about the toxic ingredients in cigarettes. Each station includes a quiz to complete by each group of students. At the end of the parcours, a moderator will announce which group of students accumulated the most points. For more information on the contents of the parcours see http://www.karuna-prevents.de/index.php.
  Arms: Student-intervention only group
Behavioral: Multi-component Intervention — One visit to the smoking prevention parcours offered by KARUNA e.V. ("Rauchst Du noch oder lebst Du schon?") + one parent night with information about smoking prevention and one informational letter by mail
  Arms: Multi-component intervention
Behavioral: Control Group — One visit to the Nutrition and Physical Activity Parcours offered by KARUNA e.V. ("Kinderleicht gesund zu leben").
  (same set up as the smoking prevention parcours with topics around healthy nutrition and promotion of physical activity)
  Arms: Control Group

SUMMARY:
The purpose of this study is to evaluate the effectiveness of a combined parent-student program for smoking prevention in 7th graders in Berlin schools.

DETAILED DESCRIPTION:
The hazardous health effects of smoking and second hand smoke are well known and published. Despite wide spread tobacco prevention campaigns and initiatives, the proportion of children and adolescents who smoke remains high, especially in Germany. Current research indicates that comprehensive strategies, especially with a parental involvement component, appear to be the most effective school-based smoking prevention programs.

A popular smoking prevention program in the city of Berlin is the Karuna interactive show jumping course "Still smoking or already alive?" ("Rauchst du noch oder lebst du schon?" Mitmach - Parcours). This parcours was designed to teach facts about smoking and its health-damaging effects, its negative effects on physical appearance, to promote communication and to enhance participants' awareness of social pressure and their self-efficacy to deal with these situations. No study to date has evaluated its effectiveness in reducing smoking rates among participating students. The study aim is to test the effectiveness of an interactive combined student-parent intervention in 7th graders regarding the reduction of smoking rates among secondary school children aged 12-15 compared to no smoking prevention intervention using self-reported questionnaires. In addition, it will be tested whether the program that involves the combination of a student and a parent intervention is more effective in the reduction of smoking rates in comparison to a program without a parental intervention.

ELIGIBILITY:
School Inclusion Criteria A school is eligible for the study if

* it is located in Berlin
* has 7th grade classes (students between 12-15 years)

School Exclusion Criteria:

* schools offers an extensive smoking prevention program for their students that includes parental involvement.
* schools that do not agree to stop visiting the KARUNA e.V. smoking parcours (if they do) for the next two years in case of being randomized to the control group.
* schools that do not agree to have a parents' night (separate or part of the typical parents' nights) where trained health coaches will introduce and discuss the topic of smoking prevention in youth in case of being randomized to the combined student-parent intervention.

Student Inclusion Criteria A student is eligible for the study if

* Female or male in the 7th grade
* Signed written assent
* Intellectual and physical ability of participant to make an informed decision about study participation
* Attends one of the participating schools
* Has signed approval from parent/caregiver

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 3400 (Estimated)
Dates: Start 2010-10; Primary Completion 2013-08 (Estimated); Study Completion 2013-08 (Estimated)

PRIMARY OUTCOMES:
Percentage of regular smokers among students at the 2 year follow-up assessment. | 2 years
  The primary study outcome is the percentage of regular smokers among students at the 2 year follow-up assessment.

SECONDARY OUTCOMES:
Students' attitudes towards smoking and smoking-related self-efficacy | 2 years
  The secondary study outcomes are attitudes towards smoking and smoking-related self-efficacy.
  In addition, we will assess the acceptability of the program components.
  Other secondary outcomes include:
  1. Percentage of 7th graders that started smoking during the study period.
  2. Percentage of 7th graders that stopped smoking during the study period.
  3. Percentage of 7th graders that are smoking less at the 2 year assessment compared to baseline assessment.
  4. Percentage of 7th graders that are smoking more at the 2 year assessment compared to baseline assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Stefan N Willich, MD, Principal Investigator — Charité University Medical Center, Institute for Social Medicine, Epidemiology and Health Economics
Locations (1):
- Charité University Medical Center, Institute for Social Medicine, Epidemiology and Health Economics, Berlin, Germany

REFERENCES:
- [Derived] Krist L, Lotz F, Burger C, Strobele-Benschop N, Roll S, Rieckmann N, Muller-Nordhorn J, Willich SN, Muller-Riemenschneider F. Long-term effectiveness of a combined student-parent and a student-only smoking prevention intervention among 7th grade school children in Berlin, Germany. Addiction. 2016 Dec;111(12):2219-2229. doi: 10.1111/add.13537. Epub 2016 Sep 19. PMID 27447693
- [Derived] Muller-Riemenschneider F, Krist L, Burger C, Strobele-Benschop N, Roll S, Rieckmann N, Muller-Nordhorn J, Willich SN. Berlin evaluates school tobacco prevention - BEST prevention: study design and methodology. BMC Public Health. 2014 Aug 23;14:871. doi: 10.1186/1471-2458-14-871. PMID 25150368